CLINICAL TRIAL: NCT03796026
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, 2-period, Crossover, Sleep Laboratory Study to Assess the Effect of Seltorexant Compared to Placebo on Respiration During Sleep in Adult Patients With Obstructive Sleep Apnea
Brief Title: A Study to Assess the Effect of Seltorexant Compared to Placebo on Respiration During Sleep in Adult Participants With Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108576; 42847922MDD1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seltorexant Followed by Placebo (Experimental): Participants will receive seltorexant (40 milligram [mg] capsules) once daily for 4 consecutive days, and after a washout period of 7 to 10 days, participants will receive matching placebo orally once daily for 4 consecutive days.
  Interventions: Drug: Seltorexant 40 mg; Drug: Placebo
- Placebo Followed by Seltorexant (Experimental): Participants will receive placebo once daily for 4 consecutive days, and after a washout period of 7 to 10 days, participants will receive seltorexant (40 mg capsules) orally once daily for 4 consecutive days.
  Interventions: Drug: Seltorexant 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: Seltorexant 40 mg — Seltorexant 40 mg capsules (over-encapsulated tablets) will be administered orally.
  Other Names: JNJ-42847922
Drug: Placebo — Matching placebo to seltorexant 40 mg capsules (over-encapsulated tablets) will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the effect of multiple doses of seltorexant compared with placebo on respiration during sleep in adult participants with mild to moderate obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a women of non-childbearing potential (WONCBP) or man. A WONCBP is defined as: a) Postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; b) Permanently sterile (permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy
* Meet the International Classification of Sleep Disorder diagnostic criteria for obstructive sleep apnea (OSA) based on the investigator's assessment with or without sleep study. The OSA diagnosis can be confirmed by previous sleep studies, appropriate documentations (for example, medical records or letters from treating physicians) or documented conversation with the treating physician
* Mild to moderate OSA, defined as AHI greater than or equal to (>=)5 to less than (<)30, based on screening polysomnography (PSG)
* Body mass index (BMI) between 18 and 40 kilogram per meter square (kg/m^2) (inclusive) (BMI = weight/height^2)
* Must be otherwise healthy based on physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. If the results of the clinical laboratory tests are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities from normal to be not clinically significant or to be appropriate and reasonable for the population under study

Exclusion Criteria:

* Has a history of, or current signs and symptoms of, severe renal insufficiency (creatinine clearance <30 milliliter per minute [mL/min]); moderate to severe hepatic insufficiency (Child-Pugh Score >=7), significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic, or endocrine disorders (including uncontrolled hypo- or hyperthyroidism or diabetes mellitus). Participants with diabetes mellitus who are under good control (hemoglobin A1c [HbA1c] <= 8.5 percent [%] and fasting glucose <=140 milligram per deciliter [mg/dL] at screening) may be eligible to participate if otherwise medically healthy, and if on a stable regimen of glucose-lowering medications for at least 2 months prior to screening
* Screening PSG with oxygen (O2) saturation <=80% for >=5% of total sleep time (TST)
* Screening PSG with >=10 periodic limb movements per hour associated with an arousal
* Currently using or used within 7 days of screening a continuous positive airway pressure (CPAP), a dental appliance, or home oxygen use for OSA, or required to use any of them for the duration of the study
* Has other respiratory disorders such as chronic obstructive pulmonary disease (COPD) or asthma that need systemic and/or inhaled steroids, bronchiectasis, or emphysema, documented by history or physical examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) Score as Measured by Polysomnography (PSG) | Day 4
  AHI score is used to indicate the severity of sleep apnea. The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. The AHI values for adults are categorized as: Normal: AHI less than (<)5, Mild sleep apnea: 5 less than or equal to (<=) AHI <15, Moderate sleep apnea: 15<= AHI <30, and Severe sleep apnea: AHI greater than or equal to (>=)30.

SECONDARY OUTCOMES:
AHI Score as Measured by PSG | Day 1 (Night)
  AHI score is used to indicate the severity of sleep apnea. The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. The AHI values for adults are categorized as: Normal: AHI <5, Mild sleep apnea: 5<= AHI <15, Moderate sleep apnea: 15<= AHI <30, and Severe sleep apnea: AHI >=30.
Mean Oxygen Saturation (SpO2) During Total Sleep Time (TST) | Nights 1 and 4
  The mean SpO2 during TST on Night 4 and Night 1 will be assessed by continuous finger pulse oximetry.
Mean SpO2 During Rapid Eye Movement (REM), Non-Rapid Eye Movement (NREM), and Awake Stages | Nights 1 and 4
  The mean SpO2 during REM, NREM and awake stages of sleep will be assessed by continuous finger pulse oximetry.
Percentage of Total Sleep Time with SpO2 less than 90 percent (%), 85%, and 80% | Nights 1 and 4
  The percentage of TST with SpO2 level less than 90%, 85%, and 80% during the night, assessed by continuous finger pulse oximetry will be reported.
Mean Latency to Persistent Sleep (LPS) as Assessed by PSG | Nights 1 and 4
  LPS is a sleep parameter and will be measured by PSG during PSG screening. Elapsed time from the beginning of the PSG recording to the onset of the first 10 minutes of continuous sleep will be measured over 4 nights and the average time to sleep will be calculated.
Wake After Sleep Onset (WASO) by PSG | Nights 1 and 4
  WASO is a sleep parameter and will be measured by PSG during PSG screening. WASO is measured during overnight sleep laboratory PSG assessment and is defined as the duration of wakefulness from the onset of persistent sleep (that is, 10 consecutive minutes of sleep) over the first 6 hours of PSG assessment. The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Sleep Efficiency (SE) by PSG | Days 1, 2, 3, and 4
  SE is a sleep parameter and will be measured by PSG during PSG screening. The total sleep time divided by the total time in bed (that is, the number of minutes from the beginning of the PSG recording to the end of the recording).
Total Sleep Time (TST) | Nights 1 and 4
  TST is a sleep parameter and will be measured by PSG during PSG screening. All of the hours of non-rapid eye movement (NREM) and rapid eye movement (REM) sleep, as measured by PSG, are summed to determine the TST.
Rapid Eye Movement (REM) Sleep Latency | Nights 1 and 4
  REM sleep is a normal stage of sleep characterized by the rapid and random movement of the eyes. REM sleep latency is the time from sleep onset until first period of REM sleep. PSG recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep).
Total Duration of Rapid Eye Movement (REM) Sleep | Nights 1 and 4
  PSG recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep). It will be calculated as number of epochs scored as REM sleep divided by 2.
NREM Sleep Latency | Nights 1 and 4
  NREM sleep latency is the time from sleep onset until first period of NREM sleep. Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: NREM sleep).
Total Duration of NREM Sleep | Nights 1 and 4
  Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: NREM sleep). It will be calculated as number of epochs scored as NREM sleep divided by 2.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Baseline up to end of study (approximately up to 9 weeks)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Percentage of Participants with all Serious Adverse Events (SAEs) and Events of Special Interest | Baseline up to end of study (approximately up to 9 weeks)
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. All SAEs and events of special interest including cataplexy (sudden, transient episode of muscle weakness accompanied by conscious awareness), sleep paralysis (the experience of not being able to move, react, or speak when falling asleep/awakening), and complex, sleep-related behaviors/parasomnias such as confusional arousals, somnambulism (sleep walking), sleep terrors, bruxism (teeth grinding), sleep sex, sleep related eating disorder, sleep behavior disorder, and catathrenia (Rapid Eye Movement [REM]-associated end-inspiratory apnea/breath holding) will be reported.
Number of Participants with Clinically Significant Vital Signs Abnormalities | Baseline up to end of study (approximately up to 9 weeks)
  Number of participants with clinically significant abnormalities in the vital signs including temperature, pulse/heart rate, respiratory rate, and blood pressure will be reported.
Number of Participants with Clinically Significant Physical Examination Abnormalities | Baseline up to end of study (approximately up to 9 weeks)
  Number of participants with clinically significant abnormalities in the physical examination including examination of height, body weight, and waist circumference will be reported.
Number of Participants with Clinically Significant Electrocardiogram (ECG) Abnormalities | Baseline up to end of study (approximately up to 9 weeks)
  Number of participants with clinically significant abnormalities in the ECG will be reported.
Number of Participants with Clinically Significant Laboratory Abnormalities | Baseline up to end of study (approximately up to 9 weeks)
  Blood samples for serum chemistry, hematology, and urinalysis will be collected for clinical laboratory testing.
Number of participants with suicidal ideation measured using Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, Days 1, 2, 4, 5, and end of study (approximately 9 weeks)
  C-SSRS is a clinician rated assessment of suicidal behavior and / or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 'yes/no' items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses are listed. Worsening of suicidal ideation indicates an increase in severity of suicidal ideation from baseline.
Bond-Lader Visual Analog Scales (B-L VAS) Score | Baseline, Day 2, and Day 5
  The B-L VAS is a patient-rated scale designed to assess the current level of sedation and consists of sixteen 100-milliliter (mm) VAS anchored by antonyms (Alert-Drowsy, Lethargic-Energetic). Scores are combined to form 3 mood factors: alertness, calmness, and contentedness. The score is measured from the left to a mark made on the line by the patient and ranges from 0 (alert) to 100 (drowsy).
Next-Day Residual Effect Measured by the Karolinska Sleepiness Scale (KSS) Score | Baseline, Day 2, and Day 5
  The KSS is a patient reported assessment of level of drowsiness at the time of scale administration. This scale is focused mainly on the propensity to fall asleep and has a high validity in measuring sleepiness. It consists of a 9-point Likert scale with response options from: 1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep).
Residual Effect on a Cognitive Test Battery Evaluated by Symbol Digit Modalities Test (SDMT) | Baseline and Day 5
  The SDMT is a widely used, paper-and-pencil assessment of complex scanning and visual tracking, requiring elements of attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed. The test is viewed as a robust screening test for adult neuropsychological impairment and has been used to demonstrate worse cognitive functioning in patients with MDD. The test includes a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. Following the key, the participant is presented with randomly ordered symbols and is required to write the number corresponding to each symbol as fast as possible. The number of correct substitutions within 90 seconds is recorded by examiner-administered cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Trail Making Test Form B (TMT-B) | Baseline and Day 5
  The TMT-B measures divided attention and executive function (tracking and sequencing). The participant is instructed to draw a line to connect a set of 25 consecutively numbered and lettered circles, alternating sequentially between numbers and letters (that is, 1-A-2-B). The participant is instructed to work as quickly as possible while still maintaining accuracy. The TMT-B has acceptable reliability; reliability coefficients have typically been reported as exceeding 0.65. The TMT-B is sensitive to cognitive decline associated with MDD.
Residual Effect on Cognitive Function Measured by Hopkins Verbal Learning Test-Revised (HVLT-R) | Baseline and Day 5
  The HVLT-R, a measure of verbal learning and memory, is a 12-item word list recall test. Administration includes 3 learning trials, a delayed recall (20-minute) trial, and a 24-word recognition list (including 12 target and 12 foil words). The test administrator reads instructions and word lists aloud, and records words recalled/recognized by the participant. Three learning trials are combined to calculate a total recall score learning, delayed recall, and recognition trials.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Clinilabs, New York, New York
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency